CLINICAL TRIAL: NCT02668120
Title: Search Elevated Serum Alkaline Phosphatase as a Marker of Prenatal Intervillositis Chronic Histiocytic (IHC)
Brief Title: Search Elevated Serum Alkaline Phosphatase as a Marker of Prenatal Intervillositis Chronic Histiocytic
Acronym: IHC
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_18; 2014-A01550-47 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Chronic Histiocytosis
Keywords: chronic histiocytic intervillositis; serum alkaline phosphatase; placenta; case-control study

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases: Patients with chronic histiocytic intervillositis during pregnancy followed at University Hospital of Lille. Alkaline phosphatase assay was performed during pregnancy and is documented in the medical record. The cases are included retrospectively.
- Low-risk pregnancy: Patients with a low risk pregnancy followed at University Hospital of Lille and recruited prospectively in prenatal consultation. These patients have no pathological obstetric history.
- High-risk pregnancy: Patients with severe pregnancy complication (IUGR, Preeclampsia or Death in Utero), but without chronic intervillositis, and hospitalized in the maternal-fetal pathology department of the University Hospital of Lille. They are recruited prospectively.

SUMMARY:
Background : Chronic histiocytic intervillositis is a rare placental disease linked with poor perinatal outcome. In a recent study, a major antenatal increased alkaline phosphatase was suspected in patients affected by chronic histiocytic intervillositis. This increase may correspond to the release of alkaline phosphatase by the syncytiotrophoblaste prejudiced in this pathology.

Aim : To confirm the association between high levels of alkaline phosphatase and the occurrence of chronic histiocytic intervillositis.

DETAILED DESCRIPTION:
Single-center study of case-control comparing three groups of patients matched for gestational age at the time of sampling. The case group will be composed of patients who experienced chronic histiocytic intervillositis which an alkaline phosphatase assay is available during pregnancy (retrospective recruitment). Two control groups will be prospectively: The first will include patients whose pregnancy is low risk. The second will consist of pathological pregnancies (IUGR, Preeclampsia and Death In Utero). All patients will have a blood sample with determination of serum alkaline phosphatase activity and examination of the placenta at delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or more
* Having signed a free and informed consent
* Enjoying a social security scheme

Inclusion criteria for cases:

* Patient who gave birth at the Lille University Hospital between 2000 and 2009.
* Lesion of intervillositis chronic histiocytic (IHC) diagnosed during histological examination of the placenta.
* An alkaline phosphatase assay during pregnancy is available and has been achieved at University Hospital of Lille.
* Prior information and not opposition of the patient to the secondary use of data collected in medical file.

Inclusion criteria for low-risk pregnancy :

* No pathological obstetric history, no current pregnancy complications
* Followed antenatal clinics at the Lille University Hospital
* A gestational age corresponding to one of the cases (pairing ± 1 week)
* No chronic intervillositis after pathological examination of the placenta

Inclusion criteria for high-risk pregnancy:

* Patient hospitalized in the maternal-fetal pathology of the Lille University Hospital Service
* Presence of IUGR, Death in Utero or severe preeclampsia with fetal repercussion
* A gestational age corresponding to one of the cases (pairing ± 1 week)
* No chronic intervillositis after pathological examination of the placenta

Exclusion Criteria:

* Twin pregnancy
* Liver disease in the interrogation
* Lack of consent of the patient
* Patient not covered by a social security scheme
* Patient minor
* Patient under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient pregnant following at the Lille University Hospital. The case group will be composed of patients who experienced chronic histiocytic intervillositis. Two control groups will be prospectively: The first will include patients whose pregnancy is low risk. The second will consist of pathological pregnancies (IUGR, Preeclampsia and Death In Utero).
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-04-16 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with alkaline phosphatase levels greater than or equal to 5 times the normal | At the time of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Damien Subtil, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU,Hôpital Jeanne de Flandres, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marchaudon V, Devisme L, Petit S, Ansart-Franquet H, Vaast P, Subtil D. Chronic histiocytic intervillositis of unknown etiology: clinical features in a consecutive series of 69 cases. Placenta. 2011 Feb;32(2):140-5. doi: 10.1016/j.placenta.2010.11.021. Epub 2010 Dec 22. PMID 21183219